CLINICAL TRIAL: NCT01756573
Title: A Study of the Effect of Dexamethasone on Duration of Upper Extremity Blocks With Bupivacaine
Brief Title: Dexamethasone and Block Duration in Upper Extremity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to continue study due to time constraints
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB12-2192
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Duration of Pain Relief
Keywords: block duration; analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bupivacaine (Active Comparator): Control
  Interventions: Drug: Bupivacaine
- Bupivacaine with Dexamethasone (Experimental): Dexamethasone will be mixed with bupivacaine
  Interventions: Drug: Dexamthsone; Drug: Bupivacaine
- Intravenous Dexamethasone (Active Comparator): Dexamethasone will be given intravenously
  Interventions: Drug: Dexamthsone; Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexamthsone
  Arms: Bupivacaine with Dexamethasone; Intravenous Dexamethasone
Drug: Bupivacaine

SUMMARY:
Effect of dexamethasone on prolonging upper extremity block is well known. But it not known if the effect comes from its local effect on the nerves or from its general analgesic effect. In this study we will compare the systemic effect to its local effect to find out if there is a difference or not.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75, no contraindication to regional anesthesia,

Exclusion Criteria:

* opioid user, chronic pain conditions, peripheral neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Malik, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine: Control
  Bupivacaine
- Bupivacaine With Dexamethasone: Dexamethasone will be mixed with bupivacaine
  Dexamthsone
  Bupivacaine
- Intravenous Dexamethasone: Dexamethasone will be given intravenously
  Dexamthsone
  Bupivacaine
Period: Overall Study
Arm/Group | Bupivacaine | Bupivacaine With Dexamethasone | Intravenous Dexamethasone
Started | 3 | 1 | 1
Completed | 3 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Bupivacaine With Dexamethasone | Intravenous Dexamethasone | Total
Number analyzed (Participants) | 3 | 1 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 1 | 5
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Analgesia Duration
Time Frame: 72 hrs
Population: study terminated prematurely due to lack of resources and participation- no data collected for Outcome measures and no analysis done
Arm/Group | Bupivacaine | Bupivacaine With Dexamethasone | Intravenous Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Bupivacaine | Bupivacaine With Dexamethasone | Intravenous Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No